CLINICAL TRIAL: NCT05743686
Title: Pilot Study of the Use of an App for the Follow-up of Oral Chemotherapy in Breast Cancer Patients
Brief Title: App for Adverse Events to Oral Chemotherapy - Pilot Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Julie Lemieux (Other)
Responsible Party: Sponsor-Investigator, Julie Lemieux, Head of Clinical Research in Breast Cancer, CHU de Quebec-Universite Laval
Organization: CHU de Quebec-Universite Laval (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021-5644
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Breast Neoplasms; Chemotherapeutic Toxicity
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Application (Experimental)
  Interventions: Device: Application

INTERVENTIONS:
Device: Application — The participants will have access to an app allowing them to report their adverse effects to oral chemotherapy. Basic advices will be given and the hospital pharmacists will be warned.

SUMMARY:
In recent years, the treatment paradigm for hormone receptor positive, HER2-negative disease has shifted from "chemotherapy for visceral disease" and "hormone therapy for bone disease" to "chemotherapy only for visceral crises or endocrine resistance". In recent years, CDK4/6 inhibitors have been added to the therapeutic arsenal. A meta-analysis of clinical trials of first-line metastatic CDK4/6 inhibitors showed an improvement in progression-free survival but an increase in toxicities compared to endocrine therapy alone. Other commonly used oral therapies for breast cancer are mTOR inhibitors and capecitabine. Other oral molecules will be added to the therapeutic arsenal in the coming years (e.g. alpelisib and tucatinib), each with specific toxicities.

Newer targeted therapies given in combination with endocrine therapies for breast cancer (eg with palbociclib, everolimus, and capecitabine) pose a challenge to health care providers because they are oral drugs. For "traditional" intravenous chemotherapy, patients must go to the hospital regularly, which allows close care by a team of doctors, pharmacists and nurses dedicated to breast cancer. On the other hand, for oral agents, monitoring is less systematic. Monitoring and managing the toxicities of oral treatments becomes a challenge. Suboptimal management of side effects can compromise patients' adherence to their treatment, have a negative impact on their side effects and increase costs for the healthcare system. Systematic follow-up is therefore necessary.

In the information age, public access to the Internet is increasing and most households in the province of Quebec now have access to the Internet, either on a smart phone, tablet or computer. Recent studies have shown that having a system to "self-report" side effects could even improve the survival of cancer patients and reduce costs. Apps allow patients to take an active role in their healthcare.

With the availability of an increasing number of oral therapies, monitoring the toxicities experienced by these patients is becoming a challenge and oncology teams need tools to help them ensure patient safety. At the same time, patients clearly want more information. The potential benefits and ease of use of web interfaces and patient portals for the management of oral therapy toxicities are appealing, but there is a lack of studies on them.

ELIGIBILITY:
Inclusion Criteria:

* >=18 years of age
* metastatic breast cancer
* receiving oral chemotherapy (palbociclib, everolimus, or capecitabine)
* possess an smartphone, a tablet, or a personal compiter

Exclusion Criteria:

* cognitive impairments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of calls | 3 months
  The number of calls to the pharmacists and the navigator nurses will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- St-Sacrement Hospital, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No